CLINICAL TRIAL: NCT07087119
Title: A Pilot Study: Exploring The Role Of an Artificial Intelligence Powered Mental Health Support Tool For Mental Health Wellness For Physicians In Training
Brief Title: Artificial Intelligence Powered Mental Health Support Tool For Physicians In Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kavya Reddy, Associate Program Director Gastroenterology Fellowship Director Adult Care Clinic Gastroenterology Assistant Clinical Professor, David Geffen School of Medicine at UCLA, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003196
Record Dates: First submitted 2025-06-09; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Wellness, Psychological; Mental Health Wellness 1
Keywords: artificial intelligence; physician in training; mental health; wellness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Masking Description: Primary Investigator and outcomes assessors will not be aware of participant information. There will only be two investigators with access to participant involvement for privacy given nature of the study. The investigators with access to participant involvement are only in place for participant safety should they need immediate help during the study. Participants will be aware of who has their information and ability to contact should they need help. However the primary investigator and investigators involved in evaluating the data will have no access to participant information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- physicians in training will enroll with maintained privacy into just the study group (Experimental): Participants will be able to engage in artificial intelligence powered mental health support session through a web browser in private sessions
  Interventions: Behavioral: utilization of artificial intelligence powered mental health support session through a web browser

INTERVENTIONS:
Behavioral: utilization of artificial intelligence powered mental health support session through a web browser — utilization of artificial intelligence powered mental health support session with the software XAIA through a web browser for physicians in training to address symptoms related to depression and anxiety.

SUMMARY:
The purpose of this pilot study is to evaluate the acceptability of an artificial intelligence powered mental health support tool for mental health wellness amongst physicians in training.

The primary research procedures are:

The primary research procedure will be the utilization of artificial intelligence powered mental health support session through a web browser for physicians in training to address symptoms related to depression and anxiety. A pre and post intervention survey, evaluating depression symptoms with the standardized PHQ-9 questionnaire and anxiety symptoms with the standardized GAD-7 questionnaire will be conducted to assess changes in mental health wellness.

The study will enroll physicians in training, including Internal Medicine residents and Gastroenterology fellows.

The study includes at least 4 sessions. The total study duration for each subject is 3 months.

DETAILED DESCRIPTION:
This is a prospective pilot study with internal medicine residents and gastroenterology fellows to evaluate the role of AI mental health support tool as a wellness resource.

Participants will be invited via e-mail to participate in the study. The invitation e-mail will describe the study and ask that those who meet exclusion criteria do not participate in this pilot study. The e-mail will also include a file with information of the study for participants to review including how study members are blinded and the de-coding process required for participants to be contacted by a study member should they score >15 on PHQ-9 and or >10 on GAD-7. Those who choose to participate will be asked to email a study member who will send the participants a REDCap link to the consent, survey and a code to be used in the survey.

Participants will be asked to complete a set of questionnaires to evaluate their mental health and factors that contribute to mental health as well as four AI powered mental health support sessions over a four-week period. This will conclude the active phase of their participations. Participants will then be sent a questionnaire at 3 months from study initiation to complete a questionnaire evaluating their mental health and if they would be interested in additional AI powered mental health support sessions.

The questionnaires will be administered before the AI sessions and at the end of the study period to evaluate for changes in mental health scores. The questionnaires will include the validated PHQ-9 for a standardized depression score and the GAD-7 for a standardized anxiety score to evaluate symptoms related to depression and anxiety. In addition, a set of questions will focus on demographics, work and home environment to evaluate factors that may contribute to mental health prior to the AI sessions and a set of questions related to the AI sessions at the end of the study period. The questionnaire will be administered via REDCap.

The AI powered sessions will be administered via a web browser such as a computer, laptop, tablets or cellphone. Participants can complete the session in the privacy of their home or in a private location at work such as a call-room. Participants will be asked to complete one 20-minute session per week during the 4-week study period for a total of four sessions.

The AI program used will be the XAIA software program. Participants will be sent an email with the link to use the XAIA software. This includes a tutorial on how to use XAIA.

The duration of the study session is 4 weeks and total duration of the study is three months.

The study will be conducted at one site only, Cedars-Sinai or participants may conduct the sessions at the privacy of their own home.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older are included.
* Training physicians in Internal Medicine residency and Gastroenterology fellowship at Cedars Sinai.
* Study is limited to Cedars-Sinai employees who are known to speak English.

Exclusion Criteria:

* Active treatment of severe and uncontrolled anxiety or depression with a health care professional
* Unwilling and or unable to participate
* Non-English speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-21 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using Artificial Intelligence sessions as a wellness resource | 3 months
  Investigators will evaluate the percentage of participants who find the Artificial Intelligence Sessions to be easily accessible and helpful.

SECONDARY OUTCOMES:
Prevalence of depression and anxiety in training physicians | 3 months
  Determine the % of participants who have symptoms of depression and anxiety in training
Determine work-related and home-related factors that impact trainee mental health | 3 months
  Evaluate percentage of participants who have work-related and home-related factors impacting mental health

CONTACTS AND LOCATIONS:
Overall Officials: Kavya Reddy, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Participant privacy

REFERENCES:
- [Background] Collier VU, McCue JD, Markus A, Smith L. Stress in medical residency: status quo after a decade of reform? Ann Intern Med. 2002 Mar 5;136(5):384-90. doi: 10.7326/0003-4819-136-5-200203050-00011. PMID 11874311
- [Background] Guille C, Frank E, Zhao Z, Kalmbach DA, Nietert PJ, Mata DA, Sen S. Work-Family Conflict and the Sex Difference in Depression Among Training Physicians. JAMA Intern Med. 2017 Dec 1;177(12):1766-1772. doi: 10.1001/jamainternmed.2017.5138. PMID 29084311
- [Background] West CP, Tan AD, Habermann TM, Sloan JA, Shanafelt TD. Association of resident fatigue and distress with perceived medical errors. JAMA. 2009 Sep 23;302(12):1294-300. doi: 10.1001/jama.2009.1389. PMID 19773564
- [Background] Dutheil F, Aubert C, Pereira B, Dambrun M, Moustafa F, Mermillod M, Baker JS, Trousselard M, Lesage FX, Navel V. Suicide among physicians and health-care workers: A systematic review and meta-analysis. PLoS One. 2019 Dec 12;14(12):e0226361. doi: 10.1371/journal.pone.0226361. eCollection 2019. PMID 31830138

DOCUMENTS (1):
  • Study Protocol (2025-06-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT07087119/Prot_000.pdf